CLINICAL TRIAL: NCT06772753
Title: Investigation of Psychedelic Effects in Psychoactive Substances
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00376501
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Psychedelic Effects in Healthy Volunteers
Keywords: psychedelic; psychoactive; healthy
MeSH Terms: interventions — Psilocybin; Ketamine; Dextromethorphan; N,N-Dimethyltryptamine; N-Methyl-3,4-methylenedioxyamphetamine; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants may receive an inactive placebo during any one of the experimental sessions.
  Interventions: Drug: Placebo
- Psilocybin (Active Comparator): Participants may receive varying oral psychoactive doses of psilocybin (4-phosphoryloxy-N,N-dimethyltryptamine)
  Interventions: Drug: Psilocybin
- Other psychoactive drugs (Experimental): Participants may receive varying oral psychoactive doses of ketamine, dextromethorphan (DXM), N,N-dimethyltryptamine (DMT), 3,4-methylenedioxymethamphetamine (MDMA), or delta-9-tetrahydrocannabinol (THC). All dose levels will be limited to doses that have been safely administered within a single day in a laboratory context in the past.
  Interventions: Drug: Ketamine; Drug: Dextromethorphan (DXM); Drug: Dimethyltryptamine (DMT); Drug: Methylenedioxymethamphetamine (MDMA); Drug: Tetrahydrocannabinol (THC)

INTERVENTIONS:
Drug: Placebo — inactive substance
  Arms: Placebo
Drug: Psilocybin — active comparator for psychedelic effects
  Arms: Psilocybin
Drug: Ketamine — psychoactive substance
  Arms: Other psychoactive drugs
Drug: Dextromethorphan (DXM) — psychoactive substance
  Arms: Other psychoactive drugs
Drug: Dimethyltryptamine (DMT) — psychoactive substance
  Arms: Other psychoactive drugs
Drug: Methylenedioxymethamphetamine (MDMA) — psychoactive substance
  Arms: Other psychoactive drugs
Drug: Tetrahydrocannabinol (THC) — psychoactive substance
  Arms: Other psychoactive drugs

SUMMARY:
The aim of this double-blind, placebo-controlled, within-subjects study is to determine whether other psychoactive substances can produce experiences akin to those seen with classic psychedelics. Screening involves a medical and psychiatric examination, including blood draw, history and physical, interviews, and questionnaires. Eligible participants will then be asked to complete up to 6 experimental drug administration session during which the participants will potentially receive and report on the subjective effects of 6 different psychoactive substances or inactive placebo. Drug assignment for some sessions will be randomized (like flipping a count or rolling a pair of dice), and both participants and study staff will be blind to the drug condition on any given day. Participants will also complete 2 preparation sessions (4 hours total) before the first experimental session, and follow-up visits after each session to discuss and debrief on the participants subjective experience.

ELIGIBILITY:
Inclusion Criteria:

* Be 25 to 55 years old
* BMI between 18 and 34 kg/m2
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the subject does not usually consume caffeinated beverages, he or she must agree not to do so on session days
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each drug administration. Exceptions include daily use of caffeine and nicotine.
* Be healthy and psychologically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree not to take any PRN prescription medications on the mornings of the sessions unless deemed appropriate by study team.

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control (e.g. oral contraceptives, intrauterine device)
* Cardiovascular conditions-coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), or transient ischemic attack-that in the clinical opinion of the screening physician or mid-level provider would put the participant at an especially high risk for adverse effects from the study.
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally acting pharmacological effect on serotonin neurons or medications that are Monoamine oxidase (MAO) inhibitors. For individuals who have intermittent or as needed (PRN) use of such medications, sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* Use of nonprescription medications, nutritional supplements, or herbal supplements except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals
* History of meeting Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for moderate or severe substance use disorder (including alcohol use disorder, but excluding tobacco), requiring that at least one of the endorsed criteria relates to prior loss of control of substance use (e.g. consuming the substance in larger amounts and for a longer amount of time than intended; persistent desire to cut down or regulate use; unsuccessful attempts to stop use; spending a great deal of time obtaining, using, or recovering from the effects of substance use).
* Active suicidal ideation and/or behavior at time of screening.
* Psychiatric disorder that in the clinical opinion of the study team would put the participant at an especially high risk for adverse effects from the study.
* First-degree relative who meets DSM-5 criteria for a Schizophrenia Spectrum or Other Psychotic Disorder (unless disorder is Substance/Medication-Induced Psychotic Disorder or Psychotic Disorder Due to Another Medical Condition), Bipolar I Disorder, or Bipolar II disorder.
* Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
* Known allergy or prior adverse reaction to any of the study drugs judged by the investigator and/or medical staff to put the study volunteer at greater risk.
* Known allergy or intolerance to nitroglycerin.
* Concomitant use of any CYP2C9 and CYP3A4 inhibitors.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mystical Experience Questionnaire (MEQ-30) | Week 2, Week 7
  The MEQ is a 30-item self-report instrument intended to assess psychedelic-specific acute subjective effects of psychoactive drugs. At the end of each experimental session, participants will be instructed to rate each of the items of the MEQ relative to the experiences that the participant encountered during the course of the drug administration session. The total score on all items is then calculated as the primary outcome measure for each experimental session.
  Scores range from 0 to 150 on this measure with higher scores reflecting more mystical experience

SECONDARY OUTCOMES:
Drug Effects Questionnaire (DEQ) | Week 2, Week 7
  The DEQ is a self-report instrument intended to assess a range of psychoactive drug effects. Individual items include ratings of abuse-related drug effects (e.g. drug effect, good effect, bad effect, liking) and behavioral/mood states often associated with drug intoxication. The DEQ will be rated at baseline prior to the first session, and then at the end of each experimental session. The the primary outcomes for each session will be DEQ score change from baseline.
  Scores range from 0 to 200 on this measure where 0 is the least impactful effect.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Barrett, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Psychedelic and Consciousness Research, Baltimore, Maryland, United States

REFERENCES:
- [Background] Strassman RJ, Qualls CR, Uhlenhuth EH, Kellner R. Dose-response study of N,N-dimethyltryptamine in humans. II. Subjective effects and preliminary results of a new rating scale. Arch Gen Psychiatry. 1994 Feb;51(2):98-108. doi: 10.1001/archpsyc.1994.03950020022002. PMID 8297217
- [Background] Ko K, Knight G, Rucker JJ, Cleare AJ. Psychedelics, Mystical Experience, and Therapeutic Efficacy: A Systematic Review. Front Psychiatry. 2022 Jul 12;13:917199. doi: 10.3389/fpsyt.2022.917199. eCollection 2022. PMID 35923458
- [Background] Schmid Y, Gasser P, Oehen P, Liechti ME. Acute subjective effects in LSD- and MDMA-assisted psychotherapy. J Psychopharmacol. 2021 Apr;35(4):362-374. doi: 10.1177/0269881120959604. Epub 2020 Oct 8. PMID 33853422
- [Background] Breeksema JJ, Niemeijer A, Kuin B, Veraart J, Vermetten E, Kamphuis J, van den Brink W, Schoevers R. Phenomenology and therapeutic potential of patient experiences during oral esketamine treatment for treatment-resistant depression: an interpretative phenomenological study. Psychopharmacology (Berl). 2023 Jul;240(7):1547-1560. doi: 10.1007/s00213-023-06388-6. Epub 2023 May 24. PMID 37222753
- [Background] Wolinsky D, Barrett FS, Vandrey R. The psychedelic effects of cannabis: A review of the literature. J Psychopharmacol. 2024 Jan;38(1):49-55. doi: 10.1177/02698811231209194. Epub 2023 Nov 10. PMID 37947321
- [Background] Earleywine M, Ueno LF, Mian MN, Altman BR. Cannabis-induced oceanic boundlessness. J Psychopharmacol. 2021 Jul;35(7):841-847. doi: 10.1177/0269881121997099. Epub 2021 Mar 28. PMID 33779383
- [Background] Reissig CJ, Carter LP, Johnson MW, Mintzer MZ, Klinedinst MA, Griffiths RR. High doses of dextromethorphan, an NMDA antagonist, produce effects similar to classic hallucinogens. Psychopharmacology (Berl). 2012 Sep;223(1):1-15. doi: 10.1007/s00213-012-2680-6. Epub 2012 Apr 13. PMID 22526529
- [Background] Carbonaro TM, Johnson MW, Hurwitz E, Griffiths RR. Double-blind comparison of the two hallucinogens psilocybin and dextromethorphan: similarities and differences in subjective experiences. Psychopharmacology (Berl). 2018 Feb;235(2):521-534. doi: 10.1007/s00213-017-4769-4. Epub 2017 Nov 7. PMID 29116367
- [Background] Barrett FS, Johnson MW, Griffiths RR. Validation of the revised Mystical Experience Questionnaire in experimental sessions with psilocybin. J Psychopharmacol. 2015 Nov;29(11):1182-90. doi: 10.1177/0269881115609019. Epub 2015 Oct 6. PMID 26442957
- [Background] Barrett FS, Griffiths RR. Classic Hallucinogens and Mystical Experiences: Phenomenology and Neural Correlates. Curr Top Behav Neurosci. 2018;36:393-430. doi: 10.1007/7854_2017_474. PMID 28401522
- [Background] Griffiths RR, Johnson MW, Richards WA, Richards BD, McCann U, Jesse R. Psilocybin occasioned mystical-type experiences: immediate and persisting dose-related effects. Psychopharmacology (Berl). 2011 Dec;218(4):649-65. doi: 10.1007/s00213-011-2358-5. Epub 2011 Jun 15. PMID 21674151